CLINICAL TRIAL: NCT01557673
Title: Effects of Bolus and Continuous Nasogastric Feeding on Small Bowel Water Content and Blood Flow
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Nottingham (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: H062011
Record Dates: First submitted 2012-03-12; First posted 2012-03-19 (Estimated); Last update posted 2013-05-06 (Estimated); Status verified 2013-05

CONDITIONS: Enteral Feeding; Nasogastric Feeding; Diarrhoea
Keywords: Nasogastric; Small bowel water; Diarrhoea; Mesenteric blood flow; Enteral feeding
MeSH Terms: conditions — Diarrhea

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- NG bolus feeding over 5 min (Active Comparator): Tube bolus (TB): feed administered via syringe through NG tube over 5 min.
  Interventions: Dietary Supplement: NG bolus feeding over 5 min
- Continuous NG feeding over 4 h (Placebo Comparator): Continuous tube drip feeding (TD): feed pump delivered via the NG tube over 4 h.
  Interventions: Dietary Supplement: Continuous NG feeding over 4 h

INTERVENTIONS:
Dietary Supplement: NG bolus feeding over 5 min — Tube bolus (TB): 400 ml of Resource® Energy Vanilla nutrient drink, Societe des Produits Nestle S.A., administered via the NG tube over 5 min.
  Other Names: Resource® Energy Vanilla nutrient drink, Societe des Produits Nestle S.A
  Arms: NG bolus feeding over 5 min
Dietary Supplement: Continuous NG feeding over 4 h — Continuous tube drip feeding (TD): 400 ml of Resource® Energy Vanilla nutrient drink, Societe des Produits Nestle S.A., delivered via feeding pump through the NG tube over 4 h.
  Other Names: Resource® Energy Vanilla nutrient drink, Societe des Produits Nestle S.A
  Arms: Continuous NG feeding over 4 h

SUMMARY:
Following surgery some patients are unable to swallow. For those requiring nutritional support a tube is sometimes passed through the nose into the stomach to provide feeding. Traditionally this type of feeding is given slowly over the course of the day. However, it is thought that this mode of feeding might increase the amount of fluid entering the bowel contributing to symptoms of diarrhoea. An alternative strategy of feeding, given in larger volumes in a shorter space of time resembles normal feeding patterns and may reduce the amount of water entering the bowel.

In this study we want to use a non invasive medical imaging technique called "magnetic resonance imaging" (or MRI) to look at the volume of bowel water following these two feeding strategies in 12 healthy volunteers.

Each volunteer will have a tube inserted into the stomach via the nose and undergo the two feeding strategies at least 7 days apart. We will take repeated images using the MRI scanner to assess the bowel response and some samples of blood are required for analysis of blood sugar.

DETAILED DESCRIPTION:
1. Background. Nutritional support is often required for undernourished patients who are unable to meet daily nutritional requirements. This is often due to lack of consciousness or problems with swallowing, Nasogastric (NG) feeding is often employed to provide active enteric nutritional support. The current approach for delivering this support usually involves pump-assisted continuous feeding spread throughout the course of a day. However, this practice is far from physiological and may promote excessive secretion of fluid into the small bowel, contributing to gastrointestinal symptoms frequently experienced by NG fed patients. Rarely, continuous enteral tube feeding has been associated with small bowel ischaemia or necrosis, although this observation has almost always been made in the critically ill. Bolus feeds given in larger volumes over shorter time periods replicate the pattern of normal feeding. Consequently gastric emptying using this method is slowed and may, therefore, reduce the metabolic demand on the small intestine and prevent excessive accumulation of small bowel fluid.
2. Aims. This study aims to investigate the influence of bolus or continuous NG feeding on small bowel fluid content and superior mesenteric blood flow. Our hypothesis is that bolus NG feeding results in lower small bowel fluid secretion and a reduction in superior mesenteric artery blood flow in comparison to individuals who are bolus NG fed.
3. Experimental protocol and methods.

   This is a single-centre, cross-over study involving 12 healthy volunteers. Two studies will be undertaken for each volunteer approximately 7 days apart:
   * Tube bolus (TB): feed administered via the NG tube over 5 min.
   * Continuous tube drip feeding (TD): feed pump delivered via the NG tube over 4 h.

   The sequence of treatment allocations will be concealed to assessors until all interventions, data collection, and statistical analysis has been completed.

   Subjects will be asked to arrive at 8:30 a.m. at the Sir Peter Mansfield Magnetic Resonance 1.5T, University of Nottingham, having abstained from alcohol, caffeine-containing drinks, and any medication for at least 24 h prior to the study, as well as having fasted overnight. An 80 cm 8FR Freka (Fresenius Kabi, Runcorn, UK) fine bore nasogastric (NG) tube will be inserted into the stomach via the nose as well as a cannula in the ante cubital fossa for blood sampling. The position of the NG tube will be verified by magnetic resonance imaging (MRI). Once the tube is sited, the volunteer will be asked to sit for 5 min in order to allow the tubes to settle and the body adapt to their presence. Following NG intubation subjects will undergo baseline MRI scanning and blood sampling for glucose, insulin and PYY. Feeding will commence at time 0. Scanning and blood tests will proceed at 30 min intervals for a total of 4 h. The feed used in all studies will be 400 ml of Resource® Energy Vanilla nutrient drink (Nestle Nutrition, Société des Produits Nestlé S.A), which is typical of a standard oral supplement.

   In the TB study arm the supplement will be administered through the NG tube via syringes over 5 min; and in the TD study the feed will be administered using a pump at a rate of 100 ml/h for 4 h.
4. Measurable end points/statistical power of the study. Primary endpoint: Small bowel water content (SBWC). Secondary endpoints: Superior mesenteric artery blood flow, gastric content emptying time, plasma concentrations of glucose, insulin and peptide YY (PYY). Previous work using mannitol and glucose indicates that mean (SD) SBWC at 40 minutes postprandially after ingesting 300ml glucose was 47 (SD 15) and using n=10 we calculate we can detect a difference of 17 ml (36%) between interventions with 90% power. We plan to recruit 12 to allow for dropouts.

ELIGIBILITY:
Inclusion Criteria:

* Healthy
* Male
* Able to undergo safe magnetic resonance scanning

Exclusion Criteria:

* Female
* Chronic medical conditions
* Regular medication
* Unable to undergo safe magentic resonance scanning
* Previous abdominal surgery
* Smoking

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2012-01; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Small bowel water volume (ml) | 0-240 min
  Small bowel water content assessed by magnetic resonance imaging.

SECONDARY OUTCOMES:
Gastric emptying | 0-240 min
  Gastric volume assessed by magnetic resonance imaging.
Superior mesenteric artery blood flow | 0-240 min
  Superior mesenteric artery blood flow and velocity assessed by magnetic resonance imaging.
Peptide YY | 0-240 min
  Serum concentration of peptide YY
Insulin | 0-240 min
  Serum concentration of insulin
Glucose | 0-240 min
  Serum concentration of glucose

CONTACTS AND LOCATIONS:
Overall Officials: Abeed H Chowdhury, BSc MRCS, Principal Investigator — University of Nottingham; Tim Bowling, MD FRCP, Study Chair — Nottingham University Hospitals NHS Trust
Locations (1):
- Sir Peter Mansfield Magnetic Resonance Centre, Nottingham, Nottinghamshire, United Kingdom

REFERENCES:
- [Background] Dempsey DT, Mullen JL, Buzby GP. The link between nutritional status and clinical outcome: can nutritional intervention modify it? Am J Clin Nutr. 1988 Feb;47(2 Suppl):352-6. doi: 10.1093/ajcn/47.2.352. PMID 3124596
- [Background] Stroud M, Duncan H, Nightingale J; British Society of Gastroenterology. Guidelines for enteral feeding in adult hospital patients. Gut. 2003 Dec;52 Suppl 7(Suppl 7):vii1-vii12. doi: 10.1136/gut.52.suppl_7.vii1. No abstract available. PMID 14612488
- [Background] Keohane PP, Attrill H, Love M, Frost P, Silk DB. Relation between osmolality of diet and gastrointestinal side effects in enteral nutrition. Br Med J (Clin Res Ed). 1984 Mar 3;288(6418):678-80. doi: 10.1136/bmj.288.6418.678. PMID 6421429
- [Background] Kocan MJ, Hickisch SM. A comparison of continuous and intermittent enteral nutrition in NICU patients. J Neurosci Nurs. 1986 Dec;18(6):333-7. doi: 10.1097/01376517-198612000-00004. PMID 2949027
- [Background] Sarap AN, Sarap MD, Childers J. Small bowel necrosis in association with jejunal tube feeding. JAAPA. 2010 Nov;23(11):28, 30-2. doi: 10.1097/01720610-201011000-00006. PMID 21086887
- [Background] Melis M, Fichera A, Ferguson MK. Bowel necrosis associated with early jejunal tube feeding: A complication of postoperative enteral nutrition. Arch Surg. 2006 Jul;141(7):701-4. doi: 10.1001/archsurg.141.7.701. PMID 16847244
- [Background] Lobo DN, Hendry PO, Rodrigues G, Marciani L, Totman JJ, Wright JW, Preston T, Gowland P, Spiller RC, Fearon KC. Gastric emptying of three liquid oral preoperative metabolic preconditioning regimens measured by magnetic resonance imaging in healthy adult volunteers: a randomised double-blind, crossover study. Clin Nutr. 2009 Dec;28(6):636-41. doi: 10.1016/j.clnu.2009.05.002. Epub 2009 Jun 4. PMID 19500889
- [Background] Hoad CL, Marciani L, Foley S, Totman JJ, Wright J, Bush D, Cox EF, Campbell E, Spiller RC, Gowland PA. Non-invasive quantification of small bowel water content by MRI: a validation study. Phys Med Biol. 2007 Dec 7;52(23):6909-22. doi: 10.1088/0031-9155/52/23/009. Epub 2007 Nov 8. PMID 18029983
- [Background] Marciani L, Cox EF, Hoad CL, Pritchard S, Totman JJ, Foley S, Mistry A, Evans S, Gowland PA, Spiller RC. Postprandial changes in small bowel water content in healthy subjects and patients with irritable bowel syndrome. Gastroenterology. 2010 Feb;138(2):469-77, 477.e1. doi: 10.1053/j.gastro.2009.10.055. Epub 2009 Nov 10. PMID 19909743